CLINICAL TRIAL: NCT00094042
Title: Work and Iron Status Evaluation (WISE)
Brief Title: Work and Iron Status Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG0007; 5R01AG020909-04 (NIH)
Record Dates: First submitted 2004-10-08; First posted 2004-10-11 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2008-08

CONDITIONS: Aging
Keywords: Socioeconomic Factors; Dietary Supplementation
MeSH Terms: interventions — Iron-Dextran Complex

INTERVENTIONS:
Drug: Iron Supplement, 120mg

SUMMARY:
This project seeks to understand how changes in the health of an individual affects the economic and social prosperity of the individual, family and community. The study involves providing iron supplements to a sample of participants in Central Java Indonesia and following those respondents for three years. They are compared with a control group who do not receive the supplement.

DETAILED DESCRIPTION:
The goal of the study is to pin down the causal effect of improvements in health on the economic and social prosperity of individuals and their families. Particular attention will be paid to the dynamics underlying the effect of health on labor outcomes; older adults are more likely to experience transitions in health and economic status and so will be emphasized.

Beginning in 2002, about 4,000 households will be interviewed every four months for about 3 years. The first two waves of the survey will serve as baselines. After the second wave, households will be randomly assigned to one of two groups. Iron supplements will be provided to all members of households assigned to one of those groups. Household members in the 2nd group will receive an identical-looking placebo. Participants will take the supplements (or placebo) on a weekly basis for a year. The study will measure the effect of supplementation on the well-being of individuals and their families.

Data will be collected at the individual, household and community level. Individual level data will cover time allocation including work and participation in community activities, earnings, self-reported and physical health and cognition. All adult household members will be interviewed; questions about children will be answered by a caretaker. Data on wealth and consumption will be collected at the household level. Community resources, services and infrastructure information will be gathered along with detailed price data.

ELIGIBILITY:
Inclusion Criteria:

* Resident in village in study area in Purworejo District, Central Java, Indonesia

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16000
Dates: Start 2002-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Thomas, Principal Investigator — Department of Economics, UCLA
Locations (1):
- Purworejo District, Central Java, Indonesia

REFERENCES:
- See also: Work and Iron Status Evaluation — http://ipl.econ.duke.edu/dthomas/WISE/index.html